CLINICAL TRIAL: NCT00934102
Title: Ophthalmic Compatibility During Seven Days of Continuous Wear of Silicone Hydrogel Lenses (P/318/08/C)
Brief Title: Ophthalmic Compatibility During Seven Days of Continuous Wear of Silicone Hydrogel Lenses
Acronym: QUINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-368-C-103
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2010-12-01 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2010-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lotrafilcon A (Active Comparator): Lotrafilcon A, silicone hydrogel, spherical contact lens randomly assigned to one eye, worn on an extended wear basis.
  Interventions: Device: Lotrafilcon A contact lens
- Narafilcon A (Active Comparator): Narafilcon A, silicone hydrogel, spherical contact lens randomly assigned to one eye, worn on an extended wear basis.
  Interventions: Device: Narafilcon A contact lens
- Galyfilcon A (Active Comparator): Galyfilcon A, silicone hydrogel, spherical contact lens randomly assigned to one eye, worn on an extended wear basis.
  Interventions: Device: Galyfilcon A contact lens

INTERVENTIONS:
Device: Narafilcon A contact lens — Investigational, silicone hydrogel, spherical soft contact lens
  Arms: Narafilcon A
Device: Lotrafilcon A contact lens — Commercially marketed, silicone hydrogel, spherical soft contact lens
  Arms: Lotrafilcon A
Device: Galyfilcon A contact lens — Commercially marketed, silicone hydrogel, spherical soft contact lens
  Arms: Galyfilcon A

SUMMARY:
The purpose of this study is to assess the ophthalmic compatibility of three different silicone hydrogel lenses worn on an overnight basis for six nights.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer
* Is correctable to a visual acuity of 20/30 or better (in each eye) with their habitual vision correction
* Has had an ocular examination in the last two years
* Is a current soft (hydrogel or silicone hydrogel) contact lens wearer
* Has clear corneas and no active ocular disease
* Can be successfully fit with the lenses to be used in the study
* Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* Is pregnant or lactating
* Has undergone corneal refractive surgery
* Currently wears lenses on an extended wear basis or was on extended wear within six months prior to the study
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research: University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 57 subjects screened for the study, 11 did not start Period 1 due to personal reasons (7) and non-suitability (4). Period 1 established Day One measurements in order to monitor changes during Period 2.
Groups:
- Narafilcon A / Lotrafilcon A: Narafilcon A experimental contact lens randomly assigned to one eye, with Lotrafilcon A commercial contact lens assigned to the fellow eye for contralateral wear.
- Narafilcon A / Galyfilcon A: Narafilcon A experimental contact lens randomly assigned to one eye, with Galyfilcon A commercial contact lens assigned to the fellow eye for contralateral wear.
- Lotrafilcon A / Galyfilcon A: Lotrafilcon A commercial contact lens randomly assigned to one eye, with Galyfilcon A commercial contact lens assigned to the fellow eye for contralateral wear.
Period: Period 1, One Night of Wear
Arm/Group | Narafilcon A / Lotrafilcon A | Narafilcon A / Galyfilcon A | Lotrafilcon A / Galyfilcon A
Started | 16 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 1 | 0 | 0
Not completed — Personal Reasons | 1 | 0 | 0
Period: Period 2, 7 Days/6 Nights of Wear
Arm/Group | Narafilcon A / Lotrafilcon A | Narafilcon A / Galyfilcon A | Lotrafilcon A / Galyfilcon A
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all subjects who were screened for the study, whether or not they subsequently were dispensed.
Arm/Group | Overall
Number analyzed (Participants) | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 23.23 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Front Surface Lens Deposits
Description: Protein and lipid deposits on the contact lens surface as assessed by the investigator using a biomicroscope, which magnifies the appearance of the contact lens on the wearer's eye. Deposits were graded on a scale of 0 to 4 with 0 being none and 4 being severe.
Time Frame: Period 2, Day 6
Population: Per Protocol. Only the data from participants who completed all study visits were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Groups:
- Lotrafilcon A; Galyfilcon A: Commercially marketed, silicone hydrogel, spherical soft contact lens, worn on an extended wear basis.
- Narafilcon A: Investigational, silicone hydrogel, spherical soft contact lens, worn on an extended wear basis.
Arm/Group | Lotrafilcon A | Narafilcon A | Galyfilcon A
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (Eyes) | 30 | 30 | 30
Units on a Scale | 0.68 (0.35) | 0.78 (0.67) | 0.77 (0.61)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 3 months.
Groups:
- Narafilcon A: Experimental, silicone hydrogel, spherical soft contact lens, worn on an extended wear basis.
Arm/Group | Lotrafilcon A | Narafilcon A | Galyfilcon A
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No distribution of trial-specific information without express written permission of director.